CLINICAL TRIAL: NCT05735015
Title: Phase 2 Study of the PTH-Independent Effects of Encaleret on Mineral Homeostasis in Subjects With Post-Surgical Hypoparathyroidism (PSH)
Brief Title: Study of the PTH-independent Effects of Encaleret on Mineral Homeostasis in Subjects With Postsurgical Hypoparathyroidism (PSH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001085; 001085-D
Record Dates: First submitted 2023-02-17; First posted 2023-02-21 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08-18

CONDITIONS: Post-Surgical Hypoparathyroidism
Keywords: Hypoparathyroidism; Hypocalcemia; Post-Surgical Hypoparathyroidism; Calcilytic; Encaleret
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All participants given 5 days of encaleret twice daily
  Interventions: Drug: encaleret

INTERVENTIONS:
Drug: encaleret — Oral administration, twice a day

SUMMARY:
Background:

Parathyroid glands in the neck make a hormone that keeps blood calcium levels stable. Sometimes these glands are damaged or removed during neck surgery. This can lead to a condition called postsurgical hypoparathyroidism (PSH). People with PSH have low levels of calcium in their blood. Calcium and vitamin D pills can help them keep their blood calcium levels steady. But this can increase calcium in the urine and result in kidney problems. New treatments for PSH are needed.

Objective:

To test a drug (encaleret) in people with PSH.

Eligibility:

People aged 18 or older who have PSH.

Design:

Participants will be in the study for 6 months. They will have a screening visit and a treatment visit.

Screening will take up to 2 days. Participants will have a physical exam. They will have blood and urine tests and tests of their heart function. They will have an ultrasound of their kidneys; they will lie on a table for 15 to 30 minutes while a wand is moved over their back.

Treatment will require participants to stay in the clinic for 7 days and 6 nights. They will take the study drug (encaleret) by mouth twice a day for 5 days. They will have a small, flexible tube inserted into a vein; this will remain in place during the visit. Blood samples will be taken through the tube 4 to 9 times each day. Participants urine will be collected.

Participants will have follow-up blood tests 1 week after leaving the clinic. They will have 3 follow-up phone calls.

DETAILED DESCRIPTION:
Study Description:

This will be a single-site, proof-of-principle, open-label study to explore the PTH-independent effects of encaleret on calcium homeostasis in participants with low or undetectable PTH levels as a result of neck surgery (PSH).

Objectives:

Primary Objective:

-Evaluate the PTH-independent effects of encaleret on renal calcium handling in participants with PSH.

Secondary Objectives:

-Evaluate the ability of encaleret to normalize blood calcium while maintaining a normal urinary calcium in participants with PSH.

Tertiary/Exploratory Objectives:

* Evaluate the ability of encaleret to increase serum iPTH levels in participants with PSH.
* Evaluate the effect of encaleret on 1-alpha hydroxylase action by measuring 1,25-(OH)2 Vitamin D levels.
* Explore the dynamic effect of encaleret on blood and urinary calcium, iPTH, cAMP, 1,25-(OH)2 Vitamin D, and urinary citrate.
* Evaluate the effect of encaleret on bone turnover in participants with PSH.
* Evaluate the effect of encaleret on phosphate, magnesium, and FGF23 levels.
* Explore the effects of encaleret on 24-hour urine markers that impact stone formation
* Examine the PK of encaleret in participants with PSH and explore PK-PD interactions.
* Explore the effect of encaleret on bone and mineral homeostasis in the following sub-groups, as defined:

  * Permanent hypoparathyroidism (Cohort 1)
  * Recent hypoparathyroidism (Cohort 2)
  * "PTH-Clamp" cohort
  * "Aparathyroid" cohort
  * Hyperthyroid cohort
  * Normothyroid cohort
  * Thyroid cancer cohort

Primary Endpoint:

-Percent change in Fractional Excretion of Calcium (FECa) from baseline (Day -1) to the final day of treatment (Day 6 or the last measurement while on encaleret). FECa calculated using fasting blood levels and spot urine collection.

Secondary Endpoints:

-Proportion of participants who achieve a concomitant normal or elevated fasting blood calcium (albumin-corrected calcium>8.5 mg/dL) and a normal 24-hour urinary calcium level (<250 mg/24 hours for women, <300 mg/24 hours for men) on encaleret at any point between day 1 and day 5.

Tertiary/Exploratory Endpoints:

* Percent change in Fractional Excretion of Calcium (FECa) from baseline (Screening visit) to the final day of treatment (Day 6 or the last measurement while on encaleret). FECa calculated using fasting blood levels and spot urine collection.
* Change in blood iPTH comparing average baseline iPTH to average peak iPTH on encaleret. The average baseline iPTH will include all baseline iPTH levels from the screening visit, Day -1, and pre-dose on Day 1. The average peak iPTH will average the peak iPTH levels on every day the patient is on encaleret (days 1 to 5). An increase in iPTH will be considered clinically significant if there is an increase both by 50% AND by more than 10 pg/dL.
* Change in 1,25-(OH)2 Vitamin D on encaleret comparing the maximal level prior to receiving calcitriol (On Days 3- 5) to baseline (Average of Day 1 Pre-dose levels). Increase will be considered significant if there is an increase of more than 50%. Participants who receive calcitriol prior to Day 3 will be excluded.

Pharmacodynamic endpoints measured over 5 days of encaleret therapy:

* Blood iPTH - Absolute levels and change from baseline
* Albumin-corrected blood calcium - Absolute levels and change from baseline
* Ionized Calcium - Absolute levels and change from baseline
* Urinary calcium clearance (fractional excretion and 24-hour total excretion) - Absolute levels and change from baseline
* Serum levels of 1,25-(OH)2 Vitamin D - Absolute levels and change from baseline
* Blood intact FGF23 (iFGF23) and C-terminal FGF23 (cFGF23) - Absolute levels and change from baseline
* Urine cAMP and citrate - Absolute levels and change from baseline
* Blood bone resorption marker, collagen crosslinked C-telopeptide (CTx) - Absolute levels and change from baseline
* Blood bone formation marker, blood procollagen type 1 N-propeptide (P1NP) - Absolute levels and change from baseline

  * PK parameters such as maximum plasma concentration Cmax), time to maximum plasma concentration (tmax), apparent terminal half-life (t 1/2)
  * Change in components of urine including: supersaturation, sodium, potassium, calcium, magnesium, chloride, phosphorus, sulfate, citrate excretion, oxalate, pH, uric acid, creatinine, osmolality, ammonium, urea nitrogen, protein catabolic rate

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet the following criteria for inclusion during screening:

1. Be able to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
2. Age >= 18 years
3. Postmenopausal women are allowed to participate in this study:

   a. Women are considered postmenopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks prior to start of the study. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment, shall she be considered not of childbearing potential.
4. Body mass index (BMI) >= 18.5 to < 39 kg/m^2
5. Have a diagnosis of PSH, either permanent PSH (Cohort 1, surgery >= 12 months ago) or recent PSH (Cohort 2, surgery < 12 months ago).
6. Participants must have achieved an albumin-corrected blood calcium level of 7.8-10.2 mg/dL on conventional therapy without significant symptoms of hypocalcemia or hypercalcemia.
7. Participants being treated with thiazide diuretics may be enrolled if they are willing and able to discontinue thiazides for at least 5 half-lives prior to initiation of encaleret and remain off during the study treatment period. (5 half-lives of hydrochlorothiazide = 75 hours; chlorothiazide = 10 hours; chlorthalidone = 12.5 days). If the thiazide is being used as an antihypertensive, as opposed to use as a urine calcium-lowering drug, alternative therapy will be offered.
8. Participants being treated with strong CYP3A4 inhibitors (including clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir) may be enrolled if they are willing and able to discontinue these medications for at least 5 half-lives prior to initiation of encaleret and remain off during the study treatment period.
9. Participants being treated with magnesium or potassium citrate supplements should discontinue such treatment starting on Day -2.
10. Participants being treated with medications that have impacts on mineral metabolism which investigators believe may impact study endpoints may be enrolled if they are willing and safely able to discontinue the medication for at least 5 half-lives prior to initiation of encaleret and remain off during the study treatment period

EXCLUSION CRITERIA:

Participants who meet any of the following criteria during Screening will not be eligible to participate in the study:

1. History of treatment with any PTH analog (i.e., PTH 1-84, PTH 1-34, TransCon PTH, etc.) within the previous 3 months
2. History of prior treatment with encaleret
3. History of hypocalcemic seizure within the past 3 months
4. Blood 25-OH Vitamin D level <25 or >60 ng/mL

   1. If subject has a blood 25-OH Vitamin D level < 25 ng/mL at the screening visit, they will be prescribed cholecalciferol or ergocalciferol supplementation. Once the 25-OH Vitamin D level is >= 25 ng/mL, the subject will be eligible to continue to the treatment phase of the study.
   2. If a subject has a blood 25-OH Vitamin D level >60 ng/mL at the screening visit, their vitamin D supplementation will be adjusted. Once the 25-OH Vitamin D level is <=60 ng/mL, the subject will be eligible to continue to the treatment phase of the study.
5. Participants with hemoglobin (Hgb) lower than the lower limit of normal.

   a. If subject has a low Hgb at the screening visit due to iron, B12, or folate deficiency, they will be prescribed supplementation. Once the Hgb level within the normal range, the subject will be eligible to continue to the treatment phase of the study.
6. Abnormal laboratory values which in the opinion of the investigator, would make the subject not suitable for participation in the study
7. Estimated glomerular filtration rate (eGFR) < 50 mL/minute/1.73 m2 using CKD-EPI.
8. Insufficient hepatic function defined as one of the following:

   * Total Bilirubin > 1.5 x ULN OR
   * Aspartate transaminase (AST) > 2x ULN OR
   * Alanine transaminase (ALT) > 2x ULN
9. 12-lead resting electrocardiogram (ECG) with clinically significant abnormalities. Participants with screening QTcF (using the Frederica equation) > 450 milliseconds (ms) will not be eligible for the treatment phase of the study.

   - If a participant has a prolonged QTcF during screening due to a reversible cause of long QT (for example hypocalcemia or QT-prolonging medications), the subject may be eligible for the treatment phase of the study if the reversible cause can be addressed, and

   repeat ECG shows QTcF <=450 milliseconds.
10. Clinically significant cardiac disease including any of the following:

    * Congestive heart failure requiring treatment (NY Heart Association grade >= 2)
    * History of clinically significant cardiac arrythmias including ventricular arrhythmias, atrial fibrillation, or conduction abnormalities
    * History of unstable angina pectoris or acute myocardial infarction
11. Participants with positive hepatitis B surface antigen (HBsAg) or Hepatitis A immunoglobulin M (IgM) at the Screening Visit. Participants who are in complete remission from Hepatitis C as evidence by sensitive assay >=12 weeks after completion of HCV therapy are allowed to participate in the study. Participants with human immunodeficiency virus (HIV) infection on a stable dose of anti-retroviral therapy who have an undetectable viral load are allowed to participate in the study.
12. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum hCG laboratory test
13. Clinically significant abnormalities in thyroid function tests. This does not include participants with non-clinically significant or treated thyroid diseases (e.g. subclinical hypothyroidism, hypothyroidism on treatment, etc). Participants on TSH-suppression therapy for thyroid cancer are allowed to participate in this study regardless of TSH level.
14. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months following the discontinuation of study treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female participants on the study the vasectomized male partner should be the sole partner for that subject.
    * Combination of the following (a+c or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier method of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
15. Sexually active male participants who are unwilling to use a condom during vaginal intercourse while taking the encaleret (study drug) and for 3 months after the last dose of the study drug. Participants should not father a child during active participation in the study starting with the first encaleret dose. Condoms are not required if the subject is vasectomized or if the subject s partner is not a woman of child-bearing potential.
16. Hypersensitivity to any active substance or excipient of encaleret
17. History of drug or alcohol dependency within 12 months preceding the Screening Visit
18. Current participation in other investigational drug studies
19. Unwillingness to refrain from blood donation within 12 weeks prior to admission visit through one year after the last dose of the study drug. If subject donated blood within 12 weeks of the screening visit, they will need to wait until 12 weeks have passed since blood donation for the admission visit.
20. Participants who have a history of diseases of mineral metabolism other than hypoparathyroidism or hyperparathyroidism which investigators believe may impact study endpoints (for example, X-linked hypophosphatemia, rickets, etc).
21. Participants with history of the following:

    * Any cancer except for thyroid cancer, basal cell skin cancer or squamous cell cancer in the last 5 years. Subjects with history of thyroid, basal cell or squamous cell cancers should have received definitive treatment for their malignancies prior to enrollment.
    * Skeletal malignancies
    * Bone metastases
    * Irradiation (radiotherapy) to the skeleton
    * Any other disease that increases the likelihood for osteosarcoma (ex. Paget s disease).
    * Unexplained elevations of alkaline phosphatase

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Effect of encaleret on Fractional Excretion of Calcium | 6 days
  Evaluate the ability of encaleret to decrease Fractional Excretion of Calcium comparing baseline (day -1) to the last day on encaleret.

SECONDARY OUTCOMES:
Effect of encaleret on achieving concomitant normal fasting blood calcium and a normal 24-hour urinary calcium level | 6 days
  Evaluate the ability of encaleret to normalize blood calcium and urinary calcium.

CONTACTS AND LOCATIONS:
Overall Officials: Iris R Hartley, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Per the IPD Sharing guidance provided, we will only be posting results of the study on Clinicaltrials.gov.

REFERENCES:
- [Background] Roberts MS, Gafni RI, Brillante B, Guthrie LC, Streit J, Gash D, Gelb J, Krusinska E, Brennan SC, Schepelmann M, Riccardi D, Bin Khayat ME, Ward DT, Nemeth EF, Rosskamp R, Collins MT. Treatment of Autosomal Dominant Hypocalcemia Type 1 With the Calcilytic NPSP795 (SHP635). J Bone Miner Res. 2019 Sep;34(9):1609-1618. doi: 10.1002/jbmr.3747. Epub 2019 Jul 26. PMID 31063613
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001085-D.html